CLINICAL TRIAL: NCT03546634
Title: Sero-conversion Study for a Two-dose Schedule of Sabin Strain Inactivated Poliovirus Vaccine in China
Brief Title: Sero-conversion Study for a Two-dose Schedule of Sabin IPV in China
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention, China (Other Government)
Collaborators: Shandong Province Centers for Disease Control and Prevention (Other)
Responsible Party: Principal Investigator, AN Zhijie, Director of Vaccine Evaluation Division, National Immunization Program, Centers for Disease Control and Prevention, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201806
Record Dates: First submitted 2018-05-23; First posted 2018-06-06 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Poliomyelitis
Keywords: Inactivated Poliovirus Vaccine; Sabin strain
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three-dose schedule for Sabin IPV (Active Comparator): Subjects vaccinate Sabin IPV at 2, 3, and 4 months of age,will be collected blood specimens twice - right before the first dose of IPV, and one month after the 3rd dose of IPV.
  Interventions: Biological: Sabin IPV
- Two-dose schedule for Sabin IPV (Experimental): Subjects first dose IPV vaccinate at 4 months of age, and the second dose IPV given between 8 and 11 months of age,will be collected blood specimens twice - right before the first dose of IPV, and one month after the 2nd dose of IPV.
  Interventions: Biological: Sabin IPV

INTERVENTIONS:
Biological: Sabin IPV — We select one Sabin IPV product, produced by China National Biotec Group, which is available for China's National Immunization Program in the selected study sites.
  Other Names: Sabin strain Inactivated Poliovirus Vaccine

SUMMARY:
This study aims to obtain the direct domestic IPV vaccine monitoring data for the CNBG products, and provide scientific evidence for the National Immunization Program and long-term polio vaccine immunization policy.

The overall objective of this research is to determine the seroconversion rates of two reduced Sabin IPV schedules in Chinese children - a 2-dose schedule and a 3-dose schedule.

DETAILED DESCRIPTION:
In April 2017, WHO/SAGE recommended that a two-dose, IPV-only schedule can be used after polio eradication, with a schedule seroconversion target of at least 90%. The recommendation was based in part on a study conducted in Cuba using Salk-IPV at 4 months and 8 months of age. However, for domestic Sabin IPVs, there are no such data to support a 2-dose schedule among Chinese infants.Two Sabin IPV products that are available to China's National Immunization Program - produced by Kunming Bio institute and China National Biotec Group (CNBG).The monitoring study on sIPV produced by Kunming Bio institute has already applied for approval.This study aims to obtain the direct domestic IPV vaccine monitoring data for the CNBG products, and provide scientific evidence for the National Immunization Program and long-term polio vaccine immunization policy.

The overall objective of this research is to determine the seroconversion rates of two reduced Sabin IPV schedules in Chinese children - a 2-dose schedule and a 3-dose schedule.

The specific objectives of the study are to:

1. Determine whether the seroconversion rate is above 90% with a 2-dose Sabin IPV schedule, with the first dose given at 4 months and the second dose given ≥4 months after the first dose.
2. Measure neutralizing antibody titers against poliovirus type I, II and III among two-dose Sabin IPV alone schedule, compared with three-dose Sabin IPV alone schedule.

ELIGIBILITY:
Inclusion Criteria:

* Parent or legal guardian agree to participate in our study.
* The family is living locally with legal residency status.

Exclusion Criteria:

* Parent or legal guardian does not agree to participate in our study.
* The potential subject has received IPV or OPV before 4 months of age in the two-dose schedule group.
* The potential subject has one or more contraindications to IPV (although we will note the contraindications).

Ages: 2 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 280 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate | 10 months
  Determine whether the seroconversion rate is above 90% using a two-dose Sabin IPV alone schedule with the first dose Sabin IPV given at 4 months and the second dose Sabin IPV given ≥4 months after the first dose.

SECONDARY OUTCOMES:
Neutralizing antibody titers | 10 months
  Measure neutralizing antibody titers against poliovirus type I, II and III among two-dose Sabin IPV-only schedules compared with three-dose Sabin IPV alone schedule.

CONTACTS AND LOCATIONS:
Overall Officials: Zijian Feng, Study Chair — Centers for Disease Control and Prevention, China
Locations (1):
- Shandong Center for Disease Control and Prevention, Jinan, China

IPD SHARING:
Plan to Share IPD: No